CLINICAL TRIAL: NCT04938895
Title: Willingness to Participate in Clinical Trials Among Black and African Americans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard University (Other)
Responsible Party: Principal Investigator, Marcella Alsan, Professor of Public Policy, Harvard University
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Health Services Research
Other Study IDs: IRB21-0864
Record Dates: First submitted 2021-06-22; First posted 2021-06-24 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Researcher-Subject Relations

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Black Woman Investigator (Experimental): Survey respondents are exposed to a Black woman investigator.
  Interventions: Behavioral: Black Respondents Exposure to a Photo
- Black Man Investigator (Experimental): Survey respondents are exposed to a Black man investigator.
  Interventions: Behavioral: Black Respondents Exposure to a Photo
- White Woman Investigator (Experimental): Survey respondents are exposed to a white woman investigator.
  Interventions: Behavioral: Black Respondents Exposure to a Photo
- White Man Investigator (Experimental): Survey respondents are exposed to a white man investigator.
  Interventions: Behavioral: Black Respondents Exposure to a Photo

INTERVENTIONS:
Behavioral: Black Respondents Exposure to a Photo — Black survey respondents will be randomly assigned to one of four treatments. In each treatment arm, the subject will view a photo of an NIH investigator. We experimentally vary treatment along two dimensions: whether the investigator is a man v. woman and whether the man is white vs. black. We will survey participants' willingness to participate in a clinical trial and how their initial response is impacted by other characteristics such as perceived trustworthiness and quality.

SUMMARY:
Despite significant racial disparities in health outcomes, racial minority groups in the United States are not adequately represented in clinical trials, and clinical trial results published in major medical journals often underreport racial demographic data of participants. Lack of diversity in clinical trials threatens the generalizability of study results and reduces the ability of minority groups to benefit from medical advancement and innovation. Prior studies show that Black men are more likely to engage in preventive services when there is racial concordance with their healthcare provider. There is minimal literature about how racial concordance or diversity in clinical trial leadership impacts study enrollment. This project examines whether patients' willingness to participate in randomized clinical trials differs based on the characteristics of the investigator.

DETAILED DESCRIPTION:
We plan to recruit subjects and randomly assign them to one of four treatments. In each treatment arm, the subject will view a photograph of a real NIH investigator. We experimentally vary treatment along two dimensions: whether the sender is Black or white and whether the sender is male or female.

Our primary aim is to assess whether the subject's stated willingness to participate in a clinical trial led by the investigator. Our secondary aim is to assess whether the subject is a more objective measure of interest in signing up for information on other clinical trials. To assess mechanisms, we will ask the respondent to rate the subject's perceived trustworthiness and quality of the investigator. In addition, we will also assess the subject's perceived attractiveness and age of the investigator as well as the subject's risk aversion, altruism, time preference, and general trust.

ELIGIBILITY:
Inclusion Criteria:

* participant identifies as Black or White

Exclusion Criteria:

* participant doesn't identify as Black or White
* younger than 25 years old, older than 64

Ages: 25 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 323 (Actual)
Dates: Start 2021-06-07 (Actual); Primary Completion 2022-02-21 (Actual); Study Completion 2022-02-21 (Actual)

PRIMARY OUTCOMES:
Willingness to Participate in a Clinical Trial | February 17, 2022 - February 19, 2022
  Survey respondents' willingness to participate in a vaccine clinical trial led by the person in the photo.

CONTACTS AND LOCATIONS:
Overall Officials: Marcella Alsan, MD,PhD, Principal Investigator — Harvard University
Locations (1):
- Harvard University, Cambridge, Massachusetts, United States